CLINICAL TRIAL: NCT00026234
Title: A Phase II Trial Evaluating Multiple Metastasectomy Combined With Hepatic Artery Infusion Of Floxuridine (FUDR) And Dexamethasone (DXM), Alternating With Systemic Oxaliplatin (OXAL) And Capecitabine (CAPCIT) For Colorectal Carcinoma Metastatic To The Liver
Brief Title: Hepatic Arterial Infusion Plus Chemotherapy in Treating Patients With Colorectal Cancer Metastatic to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01866; N9945; CDR0000069011; NCCTG-N9945; NSABP-CI-66; U10CA025224 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Liver Metastases; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Floxuridine; Dexamethasone; Calcium Dobesilate; Oxaliplatin; Capecitabine

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive floxuridine and dexamethasone intra-arterially continuously on days 1-14, oxaliplatin IV over 2 hours on day 22, and oral capecitabine twice daily on days 22-35. Treatment repeats every 6 weeks for 4 courses in the absence of disease recurrence or unacceptable toxicity. After completion of the fourth course, patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for 2 courses in the absence of disease recurrence or unacceptable toxicity.
  Interventions: Drug: floxuridine; Drug: dexamethasone; Drug: oxaliplatin; Drug: capecitabine

INTERVENTIONS:
Drug: floxuridine — Given intra-arterially
  Other Names: 5-FUDR
Drug: dexamethasone — Given intra-arterially
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda

SUMMARY:
Phase II trial to study the effectiveness of hepatic arterial infusion plus chemotherapy in treating patients who have colorectal cancer metastatic to the liver. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs in different combinations and different ways may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and toxicity of hepatic arterial infusion with floxuridine and dexamethasone followed by systemic therapy with oxaliplatin and capecitabine in patients with surgically resected liver metastases from primary colorectal carcinoma.

II. Determine the 2-year survival rate of patients treated with this regimen. III. Determine the 2-year recurrence rate and time to recurrence in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive floxuridine and dexamethasone intra-arterially continuously on days 1-14, oxaliplatin IV over 2 hours on day 22, and oral capecitabine twice daily on days 22-35. Treatment repeats every 6 weeks for 4 courses in the absence of disease recurrence or unacceptable toxicity. After completion of the fourth course, patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for 2 courses in the absence of disease recurrence or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2.5 years.

PROJECTED ACCRUAL: A total of 15-75 patients will be accrued for this study within 9 months-3.25 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma metastatic to the liver
* No extrahepatic metastases
* Prior complete surgical resection of hepatic metastases (at least 1 lesion) within the past 21-56 days

  * Negative surgical margins unless surrounding normal liver tissue was ablated during surgery
  * Radiofrequency ablation may be used as adjunct to surgical resection but not as primary treatment
  * No prior operative ultrasound during resection of hepatic metastases
* Prior complete surgical resection of carcinoma of colon or rectum (must appear completely resectable in case of synchronous lesions)
* Performance status - ECOG 0-1
* Absolute neutrophil count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* No pre-existing chronic hepatic disease (chronic active hepatitis or cirrhosis)
* Creatinine no greater than ULN
* Creatinine clearance greater than 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate oral nutrition (at least 1,500 calories/day)
* Able to withstand major operative procedure
* No dehydration
* No severe anorexia
* No frequent nausea or vomiting
* No prior or concurrent malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of any organ
* No prior or concurrent malignancy associated with more than 10% probability of death from malignant disease within 5 years of diagnosis
* No concurrent immunotherapy
* No concurrent colony-stimulating factors during the first course of study therapy
* No more than 1 prior adjuvant systemic fluorouracil (5-FU) regimen with or without levamisole, leucovorin calcium, or irinotecan

  * One prior 5-FU-based regimen as neoadjuvant treatment for rectal cancer is allowed
* No prior hepatic artery infusion therapy with 5-FU or floxuridine
* No prior systemic chemotherapy for metastatic disease
* No other concurrent chemotherapy
* No concurrent radiotherapy
* See Disease Characteristics
* No prior or concurrent sorivudine or brivudine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2002-02; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Toxicity of oxaliplatin as assessed by the National Cancer Institute (NCI) Common Terminology Criteria (CTC) version 2.0 | Up to 6 months
Survival rate | From the date of resection, cryoablation, or radiofrequency ablation to up to 2 years

SECONDARY OUTCOMES:
Survival time | Time from metastasectomy, cryoablation, or radiofrequency ablation to death due to any cause, assessed up to 3.5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to recurrence | Time from metastasectomy, cryoablation, or radiofrequency ablation to documentation of disease recurrence, assessed up to 2 years
  The distribution of the disease free interval will be estimated using the method of Kaplan-Meier.
Time to treatment failure | From the date of metastasectomy, cryoablation, radiofrequency ablation to the date at which the patient is removed from treatment due to recurrence, toxicity, or refusal, assessed up to 3.5 years
Adverse events as assessed by NCI CTC version 2.0 | Up to 3.5 years
  Patterns of treatment failure, toxicity, including complications associated with the intra-arterial catheter, will be summarized in tabular form.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Alberts, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Alberts SR, Roh MS, Mahoney MR, O'Connell MJ, Nagorney DM, Wagman L, Smyrk TC, Weiland TL, Lai LL, Schwarz RE, Molina R, Dentchev T, Bolton JS. Alternating systemic and hepatic artery infusion therapy for resected liver metastases from colorectal cancer: a North Central Cancer Treatment Group (NCCTG)/ National Surgical Adjuvant Breast and Bowel Project (NSABP) phase II intergroup trial, N9945/CI-66. J Clin Oncol. 2010 Feb 10;28(5):853-8. doi: 10.1200/JCO.2009.24.6728. Epub 2010 Jan 4. PMID 20048179